CLINICAL TRIAL: NCT02676622
Title: A Pilot Study of Autologous Hematopoietic Stem Cell Transplantation With Post-Transplant Ultra Low-Dose IL-2 for Refractory Crohn's Disease
Brief Title: Autologous Stem Cell Transplant for Refractory Crohn's Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI moved to a different institution.
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB1100448
Record Dates: First submitted 2013-04-21; First posted 2016-02-08 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Autologous Hematopoietic Stem cell Transplant; Cyclophosphamide; IL-2; Aldesleukin; Proleukin; PCDAI
MeSH Terms: conditions — Crohn Disease | interventions — Leukapheresis; Cyclophosphamide; Granulocyte Colony-Stimulating Factor; Filgrastim; Leukocyte Count; Blood Component Removal; Mesna; thymoglobulin; Stem Cell Transplantation; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem-cell mobilization and Leukapheresis (Experimental): Stem-cell mobilisation will be achieved using Cyclophosphamide (CY) 4g/m² (2g/m2 on 2 consecutive days) followed 5 days later by filgrastim (G-CSF) 10 mg/kg injection. This will be done daily until the day before the last day of leukapheresis. The PBSCs will be harvested usually between day +9 and +11 of completing CY.
  Leukapheresis will be performed to a target cell dose of 3-8 x106 CD34+ cells/kg Approximately 1 month later patients will undergo HSCT
  Interventions: Drug: mobilization of stem cells to prepare for Leukapheresis; Other: Leukapheresis- Collection of stem cells; Drug: Preparative regimen 4-6 weeks after Leukapheresis; Other: Stem Cell Transplant; Drug: Low-dose IL-2 administration

INTERVENTIONS:
Drug: mobilization of stem cells to prepare for Leukapheresis — Cyclophosphomide 2 g/m2 x 2 consecutive days.
  Filgrastim (G-csf) 10 mcg/kg SC will start 5 days after the last dose of CY and will end the day before the last leukapharesis.
  Other Names: Cytoxan; G-csf; Neupogen
Other: Leukapheresis- Collection of stem cells — Placement of an Apheresis Catheter on the day of collection of stem cells.
  Leukapheresis will be performed on a continuous flow separator machine to target 3-8 x 106 CD34+ cells/kg body weight.
  Other Names: white blood cells; Apheresis
Drug: Preparative regimen 4-6 weeks after Leukapheresis — Prior to starting medicines, a central venous line will be placed (arm or chest)
  Cyclophosphamide iv: 50 mg/kg iv over 2 hours
  Mesna iv (uro-protectant): 36 mg/kg iv over 12 hours
  r-ATG (Thymoglobulin, Genzyme): 2.5 mg/kg/dose iv over 6 hours on days -3,-2,-1
  Other Names: Cytoxan; Mesnex; Thymoglobulin; Genzyme
Other: Stem Cell Transplant — Infusion of the(cryopreserved and thawed)peripheral blood stem cells (PBSC)occurs on Day 0.
  Day +5: start Filgrastim (G-csf) subcutaneous injections
  Hospitalization in isolation room for 4-5 weeks
  Other Names: HSCT; Neupogen
Drug: Low-dose IL-2 administration — IL-2 Subcutaneous injections will start once ANC is > 500/µL and patient is afebrile (start IL-2 will be approximately day +20)for 6 weeks of treatment.
  Once patient or parent has learnt the administration and patient is tolerating it well, then the rest of the treatment can be administered at home after discharge with weekly follow up visits.
  Other Names: Aldesleukin

SUMMARY:
Crohn's disease is an 'auto-immune' disorder of the gut. In this condition the body's own immune system is fighting its gut and causing inflammation and other symptoms. Patients who are refractory (not responding) to the medications usually used to control Crohn's disease (medicines like steroids, azathioprine, methotrexate, cyclophosphamide and antibodies like Infliximab), may consider being part of this study.

In this study, the investigators plan to wipe out (ablate) the 'faulty immune system' with medicines (immune-ablation) and then give back the patients own stored stem cells (that have been collected before) - a procedure called autologous (self) stem cell transplant (ASCT). Once the new immune system regrows again from the stem cells, it is hoped that the 'faulty' immune cells do not return again and do not fight the gut leading to remission from symptoms of Crohn's disease. The aim of this treatment therefore, is to reset or re-program the immune system, so that it does not fight the patient's own body.

Currently, there are very few trials and experience with this procedure in children and young adults. There have been a few studies that have shown benefit of ASCT procedure in adult patients. In some patients, the benefit lasted for 1-5 years; but 1 in 5 (20%) participants were not taking their medications for the Crohn's disease even 5 years after ASCT. Other 80% needed medications again, but in most cases with better disease control.

In order to potentially improve the long term outcomes of ASCT, the investigators are adding another medication (in addition to those used in adult studies) called IL-2 (Aldesleukin), which will be given as an every-other-day injection under the skin (subcutaneous) at very low doses for 6 weeks after the ASCT and can be taken at home. Low dose IL-2 is known to increase a type of immune cell called T-regulatory cells (Tregs) that make immune cells less reactive to self. Study doctors believe that increased population of Tregs after ASCT may lead to a better control of Crohn's disease- higher percentage of cures or disease control for a longer period of time compared to the previous adult trials.

Therefore, the goals of this study are-

1. To see if ASCT can be used safely and can provide substantial benefit in young adults who have refractory Crohn's disease.
2. To see if addition of IL-2 after the ASCT is safe and effective.

DETAILED DESCRIPTION:
Crohn's Disease (CD) is an immunologically mediated chronic illness that has a relapsing and remitting course, most commonly presenting in the 2nd or 3rd decade and causing life long impairment of health and quality of life. Mainstay of clinical treatment for severe disease is combination of anti-inflammatory agents like 5-aminosalicyaltes and immunosuppressive medications like corticosteroids and newer anti-TNF antibodies like Infliximab. None of the drugs are, at present, curative and a relevant subset of patients are refractory to many of these pharmacologic approaches.

Immunoablative treatment followed by autologous stem cell rescue (Autologous HSCT) has been tried in this refractory group of patients with successful results. Autologous HSCT works in this auto-immune setting through the eradication of effector/memory T-cell clones due to a direct immuno-ablative effect of drugs used in the preparative regimen; by leading to an immune-reset- recovering clones of T- cells from the infused stem cells do not mount an auto-immune response and are tolerant to 'self' antigens and, by upregulation of T regulatory cells (Treg, CD4+CD25+FOXP3+ or CD8+ FOXP3+) via change in cytokine mileu during transplant. Increased population of Tregs restricts the activity of self reactive effector T-cells.

This pilot study is designed to gain on the success of previously published adult studies of autologous HSCT in refractory CD, with the aim to confirm the feasibility, safety and efficacy of HSCT and ultra low dose IL-2 when given post-HSCT in pediatric patients and young adults. IL-2 in very low doses has been shown to increase the proliferation of Treg lymphocytes and decrease inflammatory response. Hence, use of IL-2 post-transplant will result in significant and persistent increase in Treg population that may lead to more durable remissions after immunoablative therapy.

This pilot will focus on the 'safety' of this treatment in pediatric population.Since, this combination of immuno-ablative therapy followed by ultra low dose IL-2 has not been studied in children with CD, therefore transplant related mortality (TRM) and severe toxicity (> grade 3 toxicity by NCI criteria) will be monitored for 100 days post-transplant in all the patients and stopping rules will be enforced in case of excessive toxicity or TRM (>10%). Correlative studies will be performed at specific time points to assess the cytokine and inflammatory markers, immune-reconstitution and quantitative Treg cells; while clinical assessments will be done for 1 year post-HSCT for disease activity, steroid free remission period to evaluate the 'clinical efficacy' of this procedure.

The major aim of this pilot is to generate the preliminary safety and cytokine profile data to confirm the feasibility and benefit of autologous HSCT and IL-2 in children and young adults with refractory CD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 and < 30 years
* Confirmed diagnosis of Crohn's Disease -Pediatric Crohn's Disease Activity Index (PCDAI) >30 or Crohn's Disease Activity Index (CDAI) of >250 any time within 3 months prior to enrollment and any one of the following- i)Endoscopic evidence of active disease confirmed on histology within 3 months prior to enrollment, or ii) Clear evidence of active small bowel Crohn's disease on small bowel imaging within 3 months prior to enrollment.
* Refractory Crohn's Disease: Moderate to severe disease that has been unresponsive to current or prior therapy with mercaptopurine and/or azathioprine (thiopurines), methotrexate and anti-TNF therapy. Patients should have relapsing disease (i.e. > 1 exacerbation/year) or corticosteroid dependence despite current or prior thiopurines, methotrexate and anti-TNF maintenance therapy or clear demonstration of intolerance or toxicity to these drugs. Patients who fail induction therapy with corticosteroids and anti-TNF therapy, and are therefore not eligible to receive maintenance therapy with thiopurines or methotrexate will also be candidates for enrollment.
* Current active disease and problems not amenable to surgery or patient at risk for developing short bowel syndrome.
* Negative stool culture, C. difficile, and negative CMV pcr (in stool or colonic biopsy). Patients with CMV colitis will receive a trial of anti-viral treatment and only responders will be considered eligible for inclusion.
* Female patients of childbearing potential must have a documented negative serum pregnancy test within 2 weeks prior to starting the mobilization regimen.
* Patients with a prior ileostomy or colostomy may enter the study. For this group of patients', physician's global assesment will be used to assess clinical activity of CD, as Pediatric CDAI and CDAI scoring method may not be representative of disease activity.
* Patients with abscesses are eligible to enroll once the abscesses or any other significant infection has resolved.

Exclusion Criteria:

* Pregnancy or unwillingness to use adequate contraception during the study- if a woman is of childbearing age.
* HIV infection. -Organ function criteria-

  1. Renal: creatinine clearance < 50 ml/min/1.73m2 (measured or estimated).
  2. Cardiac: left ventricular ejection fraction <30% by multigated radionuclide angiography (MUGA) or a shortening fraction of < 25% by cardiac echocardiogram.
  3. Pulmonary Function tests: DLCO < 30% or patient on oxygen.
  4. Hepatic: serum bilirubin > 3 mg%; AST and ALT > 3x ULN for the institutional lab.
* Uncontrolled Hypertension (using age based criteria) despite at least 2 anti-hypertensive agents.

-Active Infection or risk thereof-

1. Current abscess or significant active infection (see 6.2.9 above)
2. Perianal infection is not an exclusion criterion, provided there is drainage with or without placement of seton.
3. Abnormal chest x ray (CXR) consistent with active infection or neoplasm.

   * Severe diarrhea due to short small bowel; pateints believed to have < 700 mm of small bowel and diarrhea attributable to this will be excluded.
   * Patients with toxic megacolon, active bowel obstruction or intestinal perforation.
   * Lack of insurance payer approval.
   * Unable to collect minimum cell dose from Leukapheresis required for transplant. These patients will be excluded from receiving the preparative regimen.

Ages: 12 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study is feasibility and safety of the autologous HSCT and low dose IL-2 post-HSCT, as evaluated by day +100 TRM (transplant related mortality) and incidence of severe toxicity. | 1 year after transplant

SECONDARY OUTCOMES:
Secondary endpoints are evaluations of the effects of HSCT on clinical and laboratory manifestations of Crohn's Disease, i.e. frequency of and types of transplant related complications that were observed. | 1 year after transplant
  Incidence of Infections: CMV reactivation and disease, adenovirus infection, BK virus reactivation, EBV PTLD and invasive fungal infections will be estimated and documented.

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Soni, MD, Principal Investigator — Nationwide Children's Hospital